CLINICAL TRIAL: NCT04835272
Title: Tracheostomy Decannulation in Severe Acquired Brain Injury: a Decannulation Protocol With Suctioning or Capping?
Brief Title: Comparison of the Decannulation Protocol With Suctioning and Capping in Severe Acquired Brain Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Song Lu, Attending doctor, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: songlu20210320
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Tracheostomy Decannulation; Acquired Brain Injury
Keywords: Tracheostomy; Decannulation; without capping; Airway patency assessment
MeSH Terms: conditions — Brain Injuries | interventions — Suction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In the control group, the decision to decannulate was based on a 48-hour capping trial.
- intervention group (Experimental): In the intervention group, the decision to decannulate was based on suctioning frequency.
  Interventions: Procedure: the Decannulation Protocol With Suctioning

INTERVENTIONS:
Procedure: the Decannulation Protocol With Suctioning — In the intervention group, the decision to decannulate was based on suctioning frequency. Patients underwent decannulation when they had had no more than two aspirations every 8 hours during during a 24-hour period. Patients in this group did not undergo capping trials.
  Other Names: the Decannulation Protocol With Capping
  Arms: intervention group

SUMMARY:
Single-center randomized trail focused on tracheostomized patients with severe acquired brain injury , comparing two different decannulation protocols:

1. an assessment of readiness for decannulation that was based on suctioning frequency
2. an assessment that was based on tracheostomy capping

ELIGIBILITY:
Inclusion Criteria:

* Within three months of onset
* Age≥18 years old
* GCS≥8
* Clinical stability( defined as the absence of fever, sepsis, or active infection and hemodynamic stability)
* Without massive pooling or silent aspiration of saliva, more than one efficient swallow per minute, adequate cough reflex were tested by gently touching the aryepiglottic region with the tip of the endoscope.
* Passing a tracheostomy-tube de-cuff test(de-cuff the tube for 3 days without pulmonary complications.
* Without significant airway stenosis.

Exclusion Criteria:

* Patients with pending diagnostic or therapeutic procedures and were considered by the clinicians to be at risk for neurologic deterioration
* Medical history of severe respiratory system or heart disease
* Neuromuscular disease other than ICU-acquired weakness, or tracheostomy for airway control
* Don't get informed consent from patient or guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
the time to decannulation | From the date of randomization to decannulation, and the patients will be followed for the duration of hospital stay, an expected average of 3 months
  the time from randomization to actual decannulation

SECONDARY OUTCOMES:
Rate of decannulation failure | within 1 week after decannulation
  reintubation within 1 week after decannulation
high dependency unit length of stay | From the date of high dependency unit admission to transferring to rehabilitation ward, and the patients will be followed for the duration of high dependency unit stay, an expected average of 2 months
  the time from high dependency unit admission to rehabilitation ward
Rate of respiratory infections | From the date of high dependency unit admission to hospital discharge, and the patients will be followed for the duration of hospital stay, an expected average of 3 months
  post decannulation respiratory infections rate in each study group
Glasgow Outcome Scale(GOS) six months after the acute brain injury | follow-up six months after discharge
  The GOS is a brief descriptive outcome scale(from 0 point to 29 points, higher score means worse outcome). GOS six months after discharge to asess the prognosis of the patient
Functional Independence Measure(FIM) six months after the acute brain injury | follow up six months after discharge
  The FIM is an 18-item ordinal scale, is viewed as most useful for assessment of progress during inpatient rehabilitation（from 18 points to 126 points, higher score means better outcome）.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wang, Study Chair — Rehabilitation medicine center, Fuxing hospital, capital medical university
Locations (1):
- Fuxing hospital, capital medical university, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication are to be shared
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after publication